CLINICAL TRIAL: NCT04129801
Title: Correlation Between Body Composition and the Muscle Strength in Severe Obese Patients in the Postoperative of Bariatric Surgery
Brief Title: Muscle Strength in Severe Obese Patients in the Postoperative of Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Roberto de Cleva, Principal investigador, University of Sao Paulo General Hospital
Other Study IDs: 01038912.6.0000.0068
Record Dates: First submitted 2019-05-21; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Severe Obesity
Keywords: Severe obesity; Body Composition; Muscle Strength; Electrical bioimpedance analysis
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective analysis: Bioimpedance The BC measurements as FM (% and kg), FFM (% and kg), will be obtained by the indirect noninvasive method of electrical bioimpedance (BIA) 230, 2.0, (Biospace Seoul, Korea). Those evaluated will be standing and positioned on the platform electrodes, barefoot and with their arms extended with their hands on the two supports (electrodes).
  Evaluation of Muscle Strength was used The Biodex Multi-joint System 3 dynamometer (Biodex Medical Systems, Inc., Shirley, New York, USA) to measure isokinetic extension (Ext) and flexion (Flex) MVC torques for both legs.
  Interventions: Other: Isokinetic Dynamometer; Other: Bioimpedance

INTERVENTIONS:
Other: Isokinetic Dynamometer — Participants then executed two series of four uninterrupted repetitions of Ext and Flex of both legs, first with the dominant member and subsequently with the non-dominant member, at an angular velocity of 60o/s, with a 60-second interval between series.
Other: Bioimpedance — Bioimpedance The BC measurements as FM (% and kg), FFM (% and kg), will be obtained by the indirect noninvasive method of electrical bioimpedance (BIA) 230, 2.0, (Biospace Seoul, Korea). Those evaluated will be standing and positioned on the platform electrodes, barefoot and with their arms extended with their hands on the two supports (electrodes).

SUMMARY:
Excessive fat mass (FM) contributes to changes in the strength and endurance of skeletal muscles. Mid-thigh muscle mass is approximately 2.5 times that of fat mass, but individuals who are obese have increased intra- (fat within muscle cells) and intermuscular fat (fat between muscle cells), establishing a negative influence on strength generation capacity and functional independence. The functional capacity of a skeletal muscle can be assessed based on the muscle's ability to produce strength. The relevance of this study is to identify/analyze the changes in segmental body composition (BC) which might better determine the association between fat free mass (FFM) of the lower limbs and maximum voluntary contraction (MVC), 36 months after bariatric surgery. This study was elaborated and will be performed at the Clinical Hospital in the Medical School of the University of Sao Paulo (HCFMUSP). The patients involved will receive the Informed Consent Form. The sample, consists of 155 adults selected at the ambulatory of the Bariatric and Metabolic Surgery Unit of the Department of Gastroenterology of HCFMUSP in the periods: preoperative, 6 and 36 months after surgery. Patients of both sexes, above 18 years of age, will undergo bariatric surgery performed at the institution. Adult patients over 60 years old, undergoing revision surgery and other surgical techniques will be excluded. Anthropometric variables will be obtained on the same day as the evaluation of BC by trained evaluators. The BC will be measured by In Body 230. BMI (kg/m2) shall be determined by dividing body weight (kg) by height (m) squared. Evaluation of Body Composition and Muscle Strength will be held between 8:00 am and 10:00 am in the Laboratory of Exercise and Movement Studies at the Institute of Orthopedics and Traumatology of FMUSP. BC measurements as FM (% and kg), FFM (% and kg), will be obtained by the indirect noninvasive method of electrical bioimpedance. The dynamometer will be used to evaluate muscle strength extension (Ext) and flexion (Flex) MVC torques for both legs will be carried. The MVC assessed variables should be absolute Ext and Flex torques (Nm), Ext and Flex torques relative to the body weight (Nm/Bw) and Ext and Flex torques relative to FFM (Nm/FFM).

DETAILED DESCRIPTION:
Anthropometric Assessment Anthropometric variables will be obtained on the same day as the evaluation of BC by trained evaluators. The body weight (kg) will be measured by In Body 230, 2.0, (Biospace Seoul, Korea). The patient should be in the orthostatic position, facing the display, in the center of the scale, barefoot, in light clothes. The height measurement (m) will be performed in a stadiometer coupled to the scale W 300, Class III, with a maximum capacity of 2m. The patient will be kept with his back to the meter, with the feet united, in an erect position, looking at horizon and arms extended to the side of the body. The reading will be made in the nearest centimeter when the horizontal rod of the vertical bar of the stature scale rests against the individual's head. BMI (kg/m2) will be determined by dividing body weight (kg) by height (m) squared.

Bioimpedance Body composition will be determined by bioelectrical impedance analysis (BIA) under constant conditions (with subjects appropriately hydrated and at the same time of day).The body composition analyzer (InBody230, Biospace Co., Gangnam-gu, Seoul, South Korea) was a segmental impedance device that uses a tetrapolar 8-point tactile electrode system, and the measured weight range was 10 to 250 kg. Impedance measurements were performed by utilizing 2 different frequencies (20 and 100 kHz) at each segment (the right arm, left arm, trunk, right leg, and left leg). The participant will be positioned in orthostatic position on a platform with lower electrodes for the feet and two brackets (the upper electrodes) gripped on hands. Data output was calculated in percentages (%) and included FM, FFM, trunk FFM, and appendicular FFM (the sum of the FFM values for the right arm, left arm, right leg, and left leg).

Isokinetic dynamometer The muscular strength evaluation will be performed on the isokinetic dynamometer, Biodex ® Multi-joint System 3 (Biodex Medical Systems Inc, Shirley, New York, USA). The dynamometer is calibrated thirty minutes before the start of the tests.

Participants are positioned for evaluation in the concentric / concentric mode of knee joint extension and flexion movements. Individuals remain seated with their hip at 90º of flexion, affixed to the chair with chest X-belts, a strap around the pelvic girdle, a strap over the distal third of the thigh and one at the distal third of the assessed leg, way to free the movements of the ankle.

All participants are instructed to perform four movements with submaximal force to familiarize themselves with the equipment. The test is performed first on the dominant limb and later on the non-dominant limb. The assessed limb is positioned with the lateral femoral condyle (axis of the knee joint movement) aligned to the mechanical axis of the dynamometer. The member that is not being evaluated will be aligned with the other member. The volunteers are instructed to perform two sets of 4 uninterrupted repetitions of knee extension and flexion with interval of 60 seconds. Throughout the period of the test, standardized and constant verbal encouragement is performed to obtain as much force as possible during contractions.

The tests are performed with concentric movements of flexion and extension of the knee, starting from 90º of flexion and reaching 20º of extension, with correction of the force of gravity.

The angular velocity used will be 60 degrees per second (60º / s).

The variables that will be obtained through the evaluation of muscular strength are:

Torque Peak (Nm): is the maximum force reached in each of the repetitions in which the test was performed. The peak torque represents the largest muscle contraction in the arc of movement and corresponds to the highest point of the force x distance curve.

Peak torque relative to body weight (Nm / kg): maximum force corrected for body weight, the result being expressed in percent newton-kilogram.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 40 and 60 kg/m2.

Exclusion Criteria:

* Functional disability
* Treatment with steroid medication for any reason.
* Use of artificial devices such as an orthosis or a prosthesis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with severe obesity undergoing bariatric surgery in the Bariatric Metabolic Surgical Unit of the Hospital das Clínicas, University of São Paulo Medical School.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Changes in Muscle strength of the lower limbs | 6 months after bariatric surgery
  Will be evaluated by Biodex Multi-joint System 3 dynamometer that measured the muscle strength of lower limbs by Extension (Ext) and flexion (Flex) torques absolute maximum voluntary contraction (MVC) Newton meter (Nm)
Changes in Muscle strength of the lower limbs | 36 months after bariatric surgery
  Will be evaluated by Biodex Multi-joint System 3 dynamometer that measured the muscle strength of lower limbs by Extension (Ext) and flexion (Flex) torques MVC, Nm
Changes in Body composition | 6 months after bariatric surgery
  Will be evaluated by electrical bioimpedance (InBody 230) that gives automatically data of: Fat Free Mass (FFM) (kg, %), Fat Mass (FM)(kg,%), Fat Free Mass of lower limbs (FFMLL) (kg, %), Fat Mass of lower limbs (FMLL) (kg,%). kilograms (Kg) e percentual (%).
Changes in Body composition | 36 months after bariatric surgery
  Will be evaluated by electrical bioimpedance (InBody 230) that gives automatically data of: FFM (kg, %), FM (kg,%), FFMLL (kg, %), FMLL (kg,%).
Changes in Muscle strength of the lower limbs relative by fat free mass of lower limbs | 6 months after bariatric surgery
  The results of muscle strength of lower limbs by Ext and Flex torques MVC Nm corrected by FFM (kg, %) obtained by assesment bioimpedance
Changes in Muscle strength of the lower limbs relative by fat free mass of lower limbs | 36 months after bariatric surgery
  The results of muscle strength of lower limbs by Ext and Flex torques MVC Nm corrected by FFM (kg, %) obtained by assesment bioimpedance
Correlate muscle strength of the lower limbs with reduction of fat free mass | 6 and 36 months after bariatric surgery
  Will be correlated the data of measured the muscle strength of lower limbs Nm with FFM (kg, %)
Correlate muscle strength of the lower limbs with reduction of fat mass | 6 and 36 months after bariatric surgery
  Will be correlated the data of measured the muscle strength of lower limbs Nm with FM (Kg, %)

SECONDARY OUTCOMES:
Muscle strength of the lower limbs relative body weight | 6 months and 36 months after bariatric surgery
  This data is obtained automatically by dynamometer that correct the muscle strength of lower limbs by body weight

CONTACTS AND LOCATIONS:
Overall Officials: Roberto de Cleva, MD Phd, Study Chair — Clinical Hospital of University of Sao Paulo Medical School; Alexandre Gadducci, MsC, Principal Investigator — University of Sao Paulo Medical School
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, Brazil

REFERENCES:
- [Background] Pereira-Lancha LO, Campos-Ferraz PL, Lancha AH Jr. Obesity: considerations about etiology, metabolism, and the use of experimental models. Diabetes Metab Syndr Obes. 2012;5:75-87. doi: 10.2147/DMSO.S25026. Epub 2012 Apr 10. PMID 22570558
- [Background] Okoro CA, Hootman JM, Strine TW, Balluz LS, Mokdad AH. Disability, arthritis, and body weight among adults 45 years and older. Obes Res. 2004 May;12(5):854-61. doi: 10.1038/oby.2004.103. PMID 15166307
- [Background] Syed IY, Davis BL. Obesity and osteoarthritis of the knee: hypotheses concerning the relationship between ground reaction forces and quadriceps fatigue in long-duration walking. Med Hypotheses. 2000 Feb;54(2):182-5. doi: 10.1054/mehy.1999.0013. PMID 10790748
- [Background] Anandacoomarasamy A, Fransen M, March L. Obesity and the musculoskeletal system. Curr Opin Rheumatol. 2009 Jan;21(1):71-7. doi: 10.1097/bor.0b013e32831bc0d7. PMID 19093327
- [Background] Hulens M, Vansant G, Claessens AL, Lysens R, Muls E. Predictors of 6-minute walk test results in lean, obese and morbidly obese women. Scand J Med Sci Sports. 2003 Apr;13(2):98-105. doi: 10.1034/j.1600-0838.2003.10273.x. PMID 12641641
- [Background] Brown M, Sinacore DR, Host HH. The relationship of strength to function in the older adult. J Gerontol A Biol Sci Med Sci. 1995 Nov;50 Spec No:55-9. doi: 10.1093/gerona/50a.special_issue.55. PMID 7493219
- [Background] Wolfson L, Judge J, Whipple R, King M. Strength is a major factor in balance, gait, and the occurrence of falls. J Gerontol A Biol Sci Med Sci. 1995 Nov;50 Spec No:64-7. doi: 10.1093/gerona/50a.special_issue.64. PMID 7493221
- [Background] Moxley Scarborough D, Krebs DE, Harris BA. Quadriceps muscle strength and dynamic stability in elderly persons. Gait Posture. 1999 Sep;10(1):10-20. doi: 10.1016/s0966-6362(99)00018-1. PMID 10469937
- [Background] Skelton DA, Kennedy J, Rutherford OM. Explosive power and asymmetry in leg muscle function in frequent fallers and non-fallers aged over 65. Age Ageing. 2002 Mar;31(2):119-25. doi: 10.1093/ageing/31.2.119. PMID 11937474
- [Background] Capodaglio P, Vismara L, Menegoni F, Baccalaro G, Galli M, Grugni G. Strength characterization of knee flexor and extensor muscles in Prader-Willi and obese patients. BMC Musculoskelet Disord. 2009 May 6;10:47. doi: 10.1186/1471-2474-10-47. PMID 19419559
- [Background] Nocera J, Buford TW, Manini TM, Naugle K, Leeuwenburgh C, Pahor M, Perri MG, Anton SD. The impact of behavioral intervention on obesity mediated declines in mobility function: implications for longevity. J Aging Res. 2011;2011:392510. doi: 10.4061/2011/392510. Epub 2011 Oct 16. PMID 22013527
- [Background] Wakeling JM, Liphardt AM, Nigg BM. Muscle activity reduces soft-tissue resonance at heel-strike during walking. J Biomech. 2003 Dec;36(12):1761-9. doi: 10.1016/s0021-9290(03)00216-1. PMID 14614930
- [Background] Taylor WR, Heller MO, Bergmann G, Duda GN. Tibio-femoral loading during human gait and stair climbing. J Orthop Res. 2004 May;22(3):625-32. doi: 10.1016/j.orthres.2003.09.003. PMID 15099644
- [Background] Gaines JM, Talbot LA. Isokinetic strength testing in research and practice. Biol Res Nurs. 1999 Jul;1(1):57-64. doi: 10.1177/109980049900100108. PMID 11225298
- [Background] Gleeson NP, Mercer TH. The utility of isokinetic dynamometry in the assessment of human muscle function. Sports Med. 1996 Jan;21(1):18-34. doi: 10.2165/00007256-199621010-00003. PMID 8771283
- [Background] O'Shea K, Kenny P, Donovan J, Condon F, McElwain JP. Outcomes following quadriceps tendon ruptures. Injury. 2002 Apr;33(3):257-60. doi: 10.1016/s0020-1383(01)00110-3. PMID 12084643
- [Background] Jaric S. Muscle strength testing: use of normalisation for body size. Sports Med. 2002;32(10):615-31. doi: 10.2165/00007256-200232100-00002. PMID 12141882
- [Background] Jaric S. Role of body size in the relation between muscle strength and movement performance. Exerc Sport Sci Rev. 2003 Jan;31(1):8-12. doi: 10.1097/00003677-200301000-00003. PMID 12562164
- [Background] De Ste Croix M, Deighan M, Armstrong N. Assessment and interpretation of isokinetic muscle strength during growth and maturation. Sports Med. 2003;33(10):727-43. doi: 10.2165/00007256-200333100-00002. PMID 12895130
- [Background] Handrigan G, Hue O, Simoneau M, Corbeil P, Marceau P, Marceau S, Tremblay A, Teasdale N. Weight loss and muscular strength affect static balance control. Int J Obes (Lond). 2010 May;34(5):936-42. doi: 10.1038/ijo.2009.300. Epub 2010 Jan 26. PMID 20101249
- [Background] Paolillo FR, Milan JC, Bueno Pde G, Paolillo AR, Borghi-Silva A, Parizotto NA, Arena R, Kurachi C, Bagnato VS. Effects of excess body mass on strength and fatigability of quadriceps in postmenopausal women. Menopause. 2012 May;19(5):556-61. doi: 10.1097/gme.0b013e3182364e80. PMID 22089183
- [Background] Koenig SM. Pulmonary complications of obesity. Am J Med Sci. 2001 Apr;321(4):249-79. doi: 10.1097/00000441-200104000-00006. PMID 11307867
- [Background] Hulens M, Vansant G, Lysens R, Claessens AL, Muls E, Brumagne S. Study of differences in peripheral muscle strength of lean versus obese women: an allometric approach. Int J Obes Relat Metab Disord. 2001 May;25(5):676-81. doi: 10.1038/sj.ijo.0801560. PMID 11360150
- [Background] Maffiuletti NA, Jubeau M, Munzinger U, Bizzini M, Agosti F, De Col A, Lafortuna CL, Sartorio A. Differences in quadriceps muscle strength and fatigue between lean and obese subjects. Eur J Appl Physiol. 2007 Sep;101(1):51-9. doi: 10.1007/s00421-007-0471-2. Epub 2007 May 3. PMID 17476522
- [Background] Gadducci AV, de Cleva R, de Faria Santarem GC, Silva PRS, Greve JMD, Santo MA. Muscle strength and body composition in severe obesity. Clinics (Sao Paulo). 2017 May;72(5):272-275. doi: 10.6061/clinics/2017(05)03. PMID 28591338
- [Background] Rolland Y, Lauwers-Cances V, Pahor M, Fillaux J, Grandjean H, Vellas B. Muscle strength in obese elderly women: effect of recreational physical activity in a cross-sectional study. Am J Clin Nutr. 2004 Apr;79(4):552-7. doi: 10.1093/ajcn/79.4.552. PMID 15051596
- [Background] Hulens M, Vansant G, Lysens R, Claessens AL, Muls E. Assessment of isokinetic muscle strength in women who are obese. J Orthop Sports Phys Ther. 2002 Jul;32(7):347-56. doi: 10.2519/jospt.2002.32.7.347. PMID 12113469
- [Background] Karelis AD, Chamberland G, Aubertin-Leheudre M, Duval C; Ecological mobility in Aging and Parkinson (EMAP) group. Validation of a portable bioelectrical impedance analyzer for the assessment of body composition. Appl Physiol Nutr Metab. 2013 Jan;38(1):27-32. doi: 10.1139/apnm-2012-0129. Epub 2013 Jan 1. PMID 23368825
- [Background] Calmels PM, Nellen M, van der Borne I, Jourdin P, Minaire P. Concentric and eccentric isokinetic assessment of flexor-extensor torque ratios at the hip, knee, and ankle in a sample population of healthy subjects. Arch Phys Med Rehabil. 1997 Nov;78(11):1224-30. doi: 10.1016/s0003-9993(97)90336-1. PMID 9365353
- [Derived] Gadducci AV, de Cleva R, Cardia L, Estabile P, Silva PRS, Greve JMD, Santo MA. Muscle Strength of Lower Limbs as a Postoperative Predictor in Bariatric Surgery. J Musculoskelet Neuronal Interact. 2024 Mar 1;24(1):31-37. PMID 38427366